CLINICAL TRIAL: NCT05745467
Title: Exploring the Impact of Nasal Povidone Iodine for Prevention of Intraoperative Spread of SARS-CoV-2 Nucleic Acid Particles and Assessment of Infectivity of Transmitted Particles
Brief Title: Povidone Iodine Nasal Application to Prevent Intraoperative Spread of SARS-CoV-2
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Wouldn't be able to get enough patients. Never started the study. Suspended the IRB form.
Sponsor: University of Iowa (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202212396
Record Dates: First submitted 2023-01-18; First posted 2023-02-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease
Keywords: General anesthetic; povidone iodine; transmission; infectivity
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Sixty-two adult patients with acute SARS-CoV-2 infection undergoing surgery (elective, urgent or emergent) at the University of Iowa will be randomized 1:1 to each of two groups, 3M 5% povidone iodine (treatment) or usual care. Vaccination status will be recorded. Patients randomized to treatment will receive 2 doses of 3M 5% nasal povidone iodine preoperatively given that this dose is commonly used to prevent surgical site infections.7 The first dose will occur prior to induction of anesthesia and the second dose will occur after induction of anesthesia and patient stabilization (in preoperative holding for elective patients or in the operating room for urgent/emergent surgery) but before incision and will involve application to each nares using 2 swabs per nares, 4 swabs per patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone Iodine (Experimental): 5% povidone iodine will be swabbed in patients' nares (experimental group), one in each nostril, twice before incision.
  Interventions: Drug: Povidone Iodine 5% Soln,Top,Kit
- Usual Care (No Intervention): Half of the patients will not receive 5% povidone iodine and will proceed with usual care.

INTERVENTIONS:
Drug: Povidone Iodine 5% Soln,Top,Kit — 5% povidone iodine will be swabbed in patients nares of the experimental group.
  Other Names: MPN: 192401; 3M Skin and Nasal Antiseptic Preoperative Preparation
  Arms: Povidone Iodine

SUMMARY:
The primary aim is to test whether preoperative asepsis with 5% nasal povidone iodine versus no preoperative asepsis with 5% nasal povidone iodine reduces proximal and distal SARS-CoV-2 transmission in operating rooms among patients who are acutely infected with SARS-CoV-2. The secondary aim is to test viral infectivity.

DETAILED DESCRIPTION:
Primary Objectives:

The primary aim is to test whether preoperative asepsis versus no preoperative asepsis reduces intraoperative SARS-CoV-2 transmission among patients acutely infected with SARS-CoV-2 (within 10 days of surgery).

Primary Endpoints:

Proximal and distal contamination with SARS-CoV-2 via nucleic acid detection.

Each patient will undergo induction of anesthesia and stabilization for the planned procedure. Approximately 50% of patients will have received 3M 5% povidone iodine 2 times prior to incision (each nares treated 2 times, 4 swabs, a total of 1 vial per patient) with the first time being before anesthesia administration and the second after anesthesia administration or usual care. Then, the investigators will sample locations for which the investigators detected SARS-CoV-2 transmission during the pilot: anesthesia work area reservoirs (anesthesia attending and assistant hands, patient nasopharynx, axilla and groin, and the anesthesia machine vaporizer at case end and at case start, and the patient intravenous stopcock at case end) and the operating room environment (anesthesia cart handles, anesthesia provider mouse, top of anesthesia cart, anesthesia suction cannister, circulating nurse mouse, walls at 6 feet, walls at the base of the floor, and air intake registers). A subset of all samples except patient nasopharynx, axilla, and groin at case beginning will be combined and processed together. Subsets of patient nasopharynx, axilla, and groin samples at case beginning will be combined and processed together. All samples will be stored separately. All samples will be collected before cleaning, transported to the laboratory, and analyzed using real-time PCR for viral detection. Samples will be saved for analysis of viral infectivity and for potential evaluation of each individual sample.

Secondary Objectives:

The secondary aim is to determine transmission of particles with infectivity.

Secondary Endpoints:

Proximal and distal environmental contamination with SARS-CoV-2 via viral culture.

All samples received in the laboratory will be assessed for infectivity in collaboration with Dr. Stanley Perlman, a preeminent expert in coronaviruses. Serial 1:10 dilutions of the 1mL primary collections in phosphate buffered saline (PBS) will be used to inoculate Vero E6 cells, incubating for 45 minutes at 37°C for plaque assay. Medium containing virus will be removed, and the cells allowed to incubate overnight in D10 media. Plaque counts will be determined the following day by combining 1% neutral red with 2× media plus agarose and incubating the cells for approximately 3 hours. All samples will be tested in triplicate with replicate experiments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Undergoing surgery (elective, urgent, or emergent)
* Requiring general anesthesia
* Acutely infected (<= 10 days from diagnosis) with SARS-CoV-2

Exclusion Criteria:

* Not general anesthesia
* Not acutely infected (<= 10 days from diagnosis) with SARS-CoV-2
* Allergy to povidone iodine
* Unable to provide consent
* Pregnant individuals

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-03 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Detection of SARS-CoV-2 nucleic acid particles in proximal and distal operating room locations using real time PCR in SARS-CoV-2 acutely infected patients receiving perioperative application of nasal 5% povidone iodine. | 4 hours
  The proximal (anesthesia attending and assistant hands, patient nasopharynx, axilla, and groin, anesthesia machine vaporizer, and patient intravenous stopcock) and distal (anesthesia cart handles, anesthesia provider mouse, top of anesthesia cart, anesthesia suction canister, circulating nurse house, walls at 6 feet and at base of the floor, and air intake registers) locations will be evaluated with real time PCR for the presence of SARS-CoV-2 nucleic acid particles. This will be evaluate for patients receiving normal care and for patients receiving nasal 5% povidone iodine preoperatively. All of the samples except for patient nasopharynx, axilla, and groin at case beginning will be pooled together and evaluated. Patient nasopharynx, axilla, and groin at case beginning will be evaluated separately.

SECONDARY OUTCOMES:
Viral load of the proximal and distal samples collected for the primary outcome will be evaluated with tissue cultures using Vero E6 cells and plaque counting. | 4 hours
  Serial 1:10 dilutions of the 1mL primary collections in phosphate buffered saline (PBS) will be used to inoculate Vero E6 cells, incubating for 45 minutes at 37°C for plaque assay. Medium containing virus will be removed, and the cells allowed to incubate overnight in D10 media. Plaque counts will be determined the following day by combining 1% neutral red with 2x media plus agarose and incubating the cells for approximately 3 hours. All samples will be tested in triplicates with replicate experiments. The amount of plaques counted will be converted into PFU/ml as the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Randy W Loftus, MD, Study Director — University of Iowa; Stephanie N Gibbons, BS, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the IPD upon review of requests. Requests will be determined appropriate or not by the PI in which the PI will decide whether or not to share the data no early than 1 year following publication of the manuscript.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will not be shared earlier than 1 year after publication of the manuscript and will be available for request for the following 2 years.
Access Criteria: I will need to determine if the request for the data is ethical and that the data will be helpful but also not used to draw false conclusions.

REFERENCES:
- [Background] Dexter F, Parra MC, Brown JR, Loftus RW. Perioperative COVID-19 Defense: An Evidence-Based Approach for Optimization of Infection Control and Operating Room Management. Anesth Analg. 2020 Jul;131(1):37-42. doi: 10.1213/ANE.0000000000004829. PMID 32217947
- [Background] Loftus RW, Dexter F, Goodheart MJ, McDonald M, Keech J, Noiseux N, Pugely A, Sharp W, Sharafuddin M, Lawrence WT, Fisher M, McGonagill P, Shanklin J, Skeete D, Tracy C, Erickson B, Granchi T, Evans L, Schmidt E, Godding J, Brenneke R, Persons D, Herber A, Yeager M, Hadder B, Brown JR. The Effect of Improving Basic Preventive Measures in the Perioperative Arena on Staphylococcus aureus Transmission and Surgical Site Infections: A Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e201934. doi: 10.1001/jamanetworkopen.2020.1934. PMID 32219407
- [Background] Loftus RW, Dexter F, Robinson ADM. High-risk Staphylococcus aureus transmission in the operating room: A call for widespread improvements in perioperative hand hygiene and patient decolonization practices. Am J Infect Control. 2018 Oct;46(10):1134-1141. doi: 10.1016/j.ajic.2018.04.211. Epub 2018 Jun 12. PMID 29907449
- [Background] Loftus RW, Dexter F, Robinson ADM. Methicillin-resistant Staphylococcus aureus has greater risk of transmission in the operating room than methicillin-sensitive S aureus. Am J Infect Control. 2018 May;46(5):520-525. doi: 10.1016/j.ajic.2017.11.002. Epub 2018 Jan 4. PMID 29307750
- [Background] Loftus RW, Dexter F, Robinson ADM, Horswill AR. Desiccation tolerance is associated with Staphylococcus aureus hypertransmissibility, resistance and infection development in the operating room. J Hosp Infect. 2018 Nov;100(3):299-308. doi: 10.1016/j.jhin.2018.06.020. Epub 2018 Jun 30. PMID 29966756
- [Background] Loftus RW, Koff MD, Brown JR, Patel HM, Jensen JT, Reddy S, Ruoff KL, Heard SO, Yeager MP, Dodds TM. The epidemiology of Staphylococcus aureus transmission in the anesthesia work area. Anesth Analg. 2015 Apr;120(4):807-18. doi: 10.1213/ANE.0b013e3182a8c16a. PMID 24937345
- [Background] Robinson ADM, Dexter F, Renkor V, Reddy S, Loftus RW. Operating room PathTrac analysis of current intraoperative Staphylococcus aureus transmission dynamics. Am J Infect Control. 2019 Oct;47(10):1240-1247. doi: 10.1016/j.ajic.2019.03.028. Epub 2019 Apr 27. PMID 31036398
- [Background] Wu S, Wang Y, Jin X, Tian J, Liu J, Mao Y. Environmental contamination by SARS-CoV-2 in a designated hospital for coronavirus disease 2019. Am J Infect Control. 2020 Aug;48(8):910-914. doi: 10.1016/j.ajic.2020.05.003. Epub 2020 May 12. PMID 32407826
- [Background] Wu J, Huang Y, Tu C, Bi C, Chen Z, Luo L, Huang M, Chen M, Tan C, Wang Z, Wang K, Liang Y, Huang J, Zheng X, Liu J. Household Transmission of SARS-CoV-2, Zhuhai, China, 2020. Clin Infect Dis. 2020 Nov 19;71(16):2099-2108. doi: 10.1093/cid/ciaa557. PMID 32392331
- [Background] Loftus RW, Dexter F, Parra MC, Brown JR. In Response: 'Perioperative COVID-19 Defense: An Evidence-Based Approach for Optimization of Infection Control and Operating Room Management'. Anesth Analg. 2020 Jul;131(1):e27-e28. doi: 10.1213/ANE.0000000000004854. No abstract available. PMID 32250978
- [Background] Chin AWH, Chu JTS, Perera MRA, Hui KPY, Yen HL, Chan MCW, Peiris M, Poon LLM. Stability of SARS-CoV-2 in different environmental conditions. Lancet Microbe. 2020 May;1(1):e10. doi: 10.1016/S2666-5247(20)30003-3. Epub 2020 Apr 2. No abstract available. PMID 32835322
- [Background] Wagner JA, Dexter F, Greeley DG, Schreiber K. Operating room air delivery design to protect patient and surgical site results in particles released at surgical table having greater concentration along walls of the room than at the instrument tray. Am J Infect Control. 2021 May;49(5):593-596. doi: 10.1016/j.ajic.2020.10.003. Epub 2020 Oct 9. PMID 33039512
- [Background] Loftus RW, Dexter F, Evans LC, Robinson ADM, Odle A, Perlman S. An assessment of the impact of recommended anesthesia work area cleaning procedures on intraoperative SARS-CoV-2 contamination, a case-series analysis. J Clin Anesth. 2021 Oct;73:110350. doi: 10.1016/j.jclinane.2021.110350. Epub 2021 May 25. No abstract available. PMID 34098391
- [Background] STONE JD, BURNET FM. The action of halogens on influenza virus with special reference to the action of iodine vapour on virus mists. Aust J Exp Biol Med Sci. 1945;23:205-12. doi: 10.1038/icb.1945.32. No abstract available. PMID 21006104